CLINICAL TRIAL: NCT03682419
Title: Evaluation of the Precision and Accuracy of International Normalised Ratio (INR) Measurements as Assessed by the LumiraDx Instrument in a Professional Point of Care Setting With Multiple Operators
Brief Title: Evaluation of Precision and Accuracy of INR Measurements in a Point of Care Device (OPTIMAL)
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D-CLIN-PROT-00001
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-09

CONDITIONS: Deep Vein Thrombosis; Atrial Fibrillation; Post-Myocardial Infarction Syndrome; Pulmonary Embolism; Artificial Heart Device User; Thrombophilia; Antiphospholipid Syndrome
MeSH Terms: conditions — Venous Thrombosis; Atrial Fibrillation; Donath-Landsteiner hemolytic anemia; Pulmonary Embolism; Thrombophilia; Antiphospholipid Syndrome

STUDY DESIGN:
Intervention Model Description: A performance evaluation study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VKA Patients (Experimental): Single Arm - blood collection by venepuncture and fingerstick in patients undergoing Warfarin Therapy
  Interventions: Procedure: VKA Patients; Procedure: Non-VKA Patients
- non-Vka Patients (Experimental): Single Arm - blood collection by venepuncture and fingerstick in patients not undergoing Warfarin Therapy
  Interventions: Procedure: VKA Patients; Procedure: Non-VKA Patients

INTERVENTIONS:
Procedure: VKA Patients — Venepuncture and capillary blood collection from Patients receiving Warfarin Therapy
  Other Names: Fingerstick to collect blood samples from Patients; Venepuncture to collect blood samples from Patients
Procedure: Non-VKA Patients — Venepuncture and capillary blood collection from Patients not receiving Warfarin Therapy
  Other Names: Fingerstick to collect blood samples from Patients; Venepuncture to collect blood samples from Patients

SUMMARY:
Comparison of capillary whole blood INR determined by LumiraDx Instrument to venous plasma INR determined by laboratory reference method (IL ACL ELITE PRO) for method comparison and assessment of accuracy and bias by regression analysis and other analytical methods.

DETAILED DESCRIPTION:
A performance evaluation study designed to assess the precision and accuracy of the LumiraDx Instrument, a point of care in vitro diagnostic system employing a portable diagnostic meter in conjunction with single use analyte test strips, for the quantitative determination of Prothrombin Time expressed as International Normalised Ratio (INR), as sampled from individuals evaluated for INR at the point of care (POC).

The accuracy of the LumiraDx Instrument INR results will be assessed by, in the first instance, comparison to the INR results obtained from the same individuals as analysed by trained laboratory professionals using the paired venous plasma samples in the reference device IL ACL ELITE PRO Coagulation Analyzer. The accuracy of INR measurements of capillary whole blood across the range of haematocrit (25% - 55%) will be assessed using paired haematocrit results obtained from the HemoCue Hb 201+ on venous whole blood. The results of these evaluations are intended to be used for regulatory filings for the LumiraDx Instrument and LumiraDx INR test as an in vitro diagnostic test in the European Union (EU) and other relevant geographies. For information only, the accuracy of the LumiraDx Instrument INR Test will also be assessed by comparison to INR results from an alternative point of care instrument, the Roche Coaguchek PRO II.

Adult males and females currently in receipt of vitamin K antagonist therapy will be included on the study. Approximately 500 subjects will be recruited to ensure that sufficient suitable subjects are enrolled and to allow for a small level of exclusions. The power calculation as well as recommendations of the FDA CLIA Waiver Guidance document (1) requires a minimum of 360 valid subjects in total (inclusive of non-therapy subset). A subsection of the subject population (~50 subjects) will consist of adult males and females who fulfil all other study inclusion criteria but are not in receipt of vitamin K antagonist therapy. This will be done in order to test the lower measurement limit of the LumiraDx Instrument INR test. At the end of the study the Healthcare Professional will be asked to complete a User Acceptability Questionnaire which is intended to assess the acceptability of the LumiraDx INR system in terms of ease of use.

ELIGIBILITY:
Inclusion Criteria - VKA Therapy Subjects:

* Persons >18 years of age
* Willing and able to provide written informed consent and comply with study procedures
* Currently prescribed vitamin K antagonist therapy
* Deemed medically appropriate for study participation by the Investigator

Exclusion Criteria - VKA Therapy Subjects:

* Persons <18 years of age
* Subject has previously participated in this study
* Subject is within 4 weeks of first prescription of vitamin K antagonist therapy
* Confirmed or suspected pregnancy
* Unwilling or unable to provide written informed consent and comply with study procedures
* Vulnerable populations deemed inappropriate for study by the Investigator
* Deemed medically inappropriate for study by the Investigator (i.e. patients with a known inherited [e.g. haemophilia or von Willebrand's disease] or acquired [e.g. liver cirrhosis] condition likely to be associated with a coagulopathy; or patients receiving non-VKA anticoagulant medications)

Inclusion Criteria - Non-VKA Therapy Subjects:

* Persons >18 years of age
* Willing and able to provide written informed consent and comply with study procedures
* Deemed medically appropriate for study participation by the Investigator

Exclusion Criteria - Non-VKA Therapy Subjects:

* Persons <18 years of age
* Subject has previously participated in this study
* Confirmed or suspected pregnancy
* Unwilling or unable to provide written informed consent and comply with study procedures
* Vulnerable populations deemed inappropriate for study by the Investigator
* Any persons deemed medically inappropriate for study by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
To determine the clinical performance of the LumiraDx instrument | 8 weeks
  Measurement of INR using Capillary & Venous blood samples

SECONDARY OUTCOMES:
To determine the accuracy of the LumiraDx instrument | 8 weeks
  Measurement of INR & Haematocrit using Capillary & Venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Tait, BSc (Hons), Principal Investigator — Consultant Haematologist
Locations (3):
- United Kingdom (3):
  - Glasgow Royal Infirmary Clinical Research Facility, Glasgow
  - Golden Jubilee National Hospital, Glasgow
  - Wishaw General Hospital, NHS Lanarkshire, Wishaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tait RC, Hung A, Gardner RS. Performance of the LumiraDx Platform INR Test in an Anticoagulation Clinic Point-of-Care Setting Compared With an Established Laboratory Reference Method. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619890423. doi: 10.1177/1076029619890423. PMID 31773973